CLINICAL TRIAL: NCT00392938
Title: Positron Emission Tomography Imaging of Bone in Patients With Metastatic Prostate Cancer - A Pilot Study Evaluating Treatment Response
Brief Title: Carbon-11 Acetate and Fludeoxyglucose F 18 PET Scan of the Bone in Patients With Metastatic Prostate Cancer That Has Spread to the Bone
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Evan Y. Yu, MD, Principal Investigator, University of Washington
Other Study IDs: 6129; P30CA015704 (NIH); UWCC-6129; UWCC-06-0500-H/A; FHCRC-6129; CDR0000480347 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Androgen Antagonists; Docetaxel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: antiandrogen therapy
Drug: docetaxel
Diagnostic Test: C-11 acetate PET scan
Diagnostic Test: F-18 FDG PET scan
Diagnostic Test: Tc-99m bone scan
Diagnostic Test: CT scan of the chest, abdomen and pelvis

SUMMARY:
RATIONALE: Imaging procedures, such as PET scan, may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This clinical trial is studying carbon-11 acetate and fludeoxyglucose F 18 PET scan of the bone in patients with metastatic prostate cancer that has spread to the bone.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Correlate pre-treatment and 3-month post-treatment carbon-11 (^11C) acetate and fludeoxyglucose F 18 positron emission tomography (^18F-FDG PET) images with changes in clinical response measures in patients with bone-dominant metastatic prostate cancer.

Secondary

* Compare ^11C acetate and ^18F-FDG PET scanning results with bone scintigraphy in these patients to determine which best predicts clinical response.
* Correlate changes in ^11C acetate and ^18F-FDG PET with changes in prostate-specific antigen level.
* Correlate changes in ^11C acetate and ^18F-FDG PET with clinical symptom parameters (pain scale scores and analgesic usage scales).
* Correlate ^11C acetate and ^18F-FDG PET scan response with clinical time to progression.
* Determine if PET scan response can predict duration of progression-free survival.

OUTLINE: This is a pilot study. Patients are stratified according to hormone response (sensitive [stratum 1] vs refractory [stratum 2]).

Patients undergo carbon-11 acetate and fludeoxyglucose F 18 positron emission tomography imaging prior to and 3 months after initiation of either androgen-deprivation therapy (stratum 1) or docetaxel (stratum 2).

Pain and quality of life are assessed at baseline and at 3 months.

Patients are followed every 3 months for up to 5 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer, meeting 1 of the following criteria:

  * Metastatic hormone-sensitive disease prior to initiation of first-line androgen-deprivation therapy and meets the following criteria:

    * Histologic confirmation of original diagnosis
    * Hormone-sensitive is defined as progressive disease in the absence of androgen-deprivation therapy
    * Presence of ≥ 3 convincing bone metastases, as defined by bone scintigraphy, CT scan (MRI if indicated), or plain x-ray
  * Metastatic hormone-refractory disease prior to initiation of a first-line chemotherapy regimen that includes docetaxel and meets the following criteria:

    * Histologic confirmation of original diagnosis
    * Hormone-refractory is defined as development or advancement of metastatic disease with castrate testosterone levels (total testosterone < 20 ng/dL)
    * Presence of ≥ 3 convincing bone metastases, as defined by bone scintigraphy, CT scan (MRI if indicated), or plain x-ray
    * Must have castrate testosterone levels (< 20 ng/dL) from orchiectomy or undergoing maintenance with a luteinizing hormone-releasing hormone agonist

      * Outside the window of a potential antiandrogen withdrawal response (either decline in prostate-specific antigen or objective response by imaging)

PATIENT CHARACTERISTICS:

* Life expectancy > 12 weeks
* No serious underlying medical condition that would otherwise impair the patient's ability to receive treatment and undergo imaging studies
* No condition that would alter the patient's mental status, prohibiting the basic understanding and/or authorization of informed consent
* Able to lie still for the imaging
* Weight ≤ 300 lbs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior bicalutamide or nilutamide
* At least 4 weeks since prior flutamide, ketoconazole, diethylstilbestrol, or estradiol
* More than 4 weeks since prior bisphosphonate therapy
* More than 4 weeks since prior radiotherapy to the bone
* More than 4 weeks since prior radiopharmaceutical treatment to the bone
* No concurrent radiotherapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-12; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Correlation of pre-treatment and 3-month post-treatment carbon-11 (11C) acetate and fludeoxyglucose F 18 positron emission tomography (18F-FDG PET) images with changes in clinical response measures

SECONDARY OUTCOMES:
Comparison of 11C acetate and 18F-FDG PET scanning results with bone scintigraphy to determine which best predicts clinical response
Correlation of changes in 11C acetate and 18F-FDG PET with changes in prostate-specific antigen level
Correlation of changes in 11C acetate and 18F-FDG PET with clinical symptom parameters (pain scale scores and analgesic usage scales)
Correlation of changes in 11C acetate and 18F-FDG PET with clinical time to progression
PET scan response as a predictor of duration of progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Evan Y. Yu, MD, Study Chair — Seattle Cancer Care Alliance
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington